CLINICAL TRIAL: NCT06554899
Title: The Efficacy of a Brief Oncologist-delivered Intervention for Fear of Cancer Recurrence: A Cluster-randomized Controlled Trial
Brief Title: CIFeR - A Clinician-led Intervention to Address Fear of Cancer Recurrence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Robert (Bobby) Zachariae, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB: R344-A19722
Record Dates: First submitted 2024-06-14; First posted 2024-08-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Fear of Cancer Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (delivering CIFeR) (Experimental): At the patient's first follow-up appointment after anti-cancer treatment, oncologists will, in addition to the usual follow-up procedure, deliver a brief psychological intervention (CIFeR)
  Interventions: Other: Clinician-led intervention to address fear of cancer recurrence (CIFeR)
- Control (treatment as usual) (No Intervention): At the patients first follow-up appointment after anti-cancer treatment, oncologists will deliver treatment as usual (the usual follow-up procedure)

INTERVENTIONS:
Other: Clinician-led intervention to address fear of cancer recurrence (CIFeR) — The intervention includes five components informed by theoretical models and existing interventions for FCR: 1) FCR normalization: reassurance that FCR is a common and normal phenomenon after treatment for cancer, 2) Providing prognostic information: asking patients whether they would like information about their risk of recurrence and, if yes,providing this information, 3) Providing education and take-home information on red-flag recurrence symptoms, 4) Brief advice on managing worry: distraction, meditation, mindfulness, reassurance, and links to online resources to manage FCR, and 5) referral to a psychologist if FCR is high (FCRI-SF >= 22), or if deemed helpful by the patient or clinician. Access will be provided to ConquerFear-Group delivered online by trained psychologists.
  Arms: Intervention (delivering CIFeR)

SUMMARY:
The investigators will test a novel Clinician-led Intervention to address Fear of cancer Recurrence in cancer survivors (CIFeR), by 1) adapting the original Australian intervention manual to the Danish oncology context (CIFeR-DK), and 2) developing a brief e-learning program to train oncologists. The investigators will then 3) compare CIFeR-DK with an active control condition in a cluster-randomized controlled trial with 24 oncologists (the cluster unit) treating a minimum of 300 patients with breast, ovarian, lung and prostate cancer at Danish Oncology Departments at four hospitals in Aarhus, Vejle, Aalborg, and Copenhagen, and 4) explore fidelity, acceptability, feasibility, and perceived barriers and facilitators to use the intervention in routine follow-up care.

DETAILED DESCRIPTION:
STUDY DESIGN:

The study is designed as a parallel cluster-randomized controlled trial with oncologists (cluster unit) treating breast, ovarian, and prostate cancer at the oncology departments at Aarhus University Hospital (AUH), Vejle Hospital (VH), Aalborg University Hospital (AAUH), and Copenhagen University Hospital (CUH), and randomized 1:1 to intervention versus active control.

Participants:

All oncologists treating breast, ovarian, and prostate cancer at the participating departments are eligible for the study and will be recruited by our collaborators at the participating departments. Eligible patients score >= 13 on the FCRI-SF and have completed their primary treatment i.e., surgery, adjuvant chemotherapy, and/or radiotherapy, for breast, ovarian, lung and prostate cancer at the participating departments between three weeks and three months previously.

Procedure:

Patients scheduled for a follow-up visit with the participating oncologists will receive a secure e-mail invitation to participate in the study and a link to a RedCap questionnaire. Patients willing to participate will provide their informed consent electronically and complete the 9-item FCRI-SF. Patients scoring >= 13 are provided with additional information about the study and asked for their consent to participate.

One week before the planned follow-up consultation, they will be asked to complete a RedCap baseline questionnaire (T1). One week and three months after the consultation, the patients will be asked to complete the RedCap post-intervention (T2) and follow-up questionnaires (T3).

Oncologists will complete a RedCap baseline questionnaire assessing age, gender, years of experience, and self-efficacy in managing patient FCR. Oncologists will then be allocated to the intervention or active control arm using a stratified randomization sequence generated by the Aarhus University clinical trial unit ensuring a balanced allocation of oncologists according to the cancer type treated. Oncologists will then receive a link to online CIFeR training and report their post-training self-efficacy for managing patient FCR. During the consultation, the oncologist will deliver the CIFeR intervention and complete a brief 5-item checklist on whether they delivered all five components and, if not, why. After including all patients, the oncologist is asked to complete a follow-up RedCap questionnaire on self-efficacy in managing patient FCR.

The CIFeR intervention:

The intervention includes five components informed by theoretical models and existing interventions for FCR: 1) FCR normalization: reassurance that FCR is a common and normal phenomenon after treatment for cancer, 2) Providing prognostic information: asking patients whether they would like information about their risk of recurrence and, if yes, providing this information, 3) Providing education and take-home information on red-flag recurrence symptoms, 4) Brief advice on managing worry: distraction, meditation, mindfulness, reassurance, and links to online resources to manage FCR, and 5) referral to a psychologist if FCR is high (FCRI-SF >= 22), or if deemed helpful by the patient or clinician. Access will be provided to ConquerFear-Group delivered online by trained psycho-oncologists.

Outcome measures:

Patients:

The primary outcome is the change in FCR, assessed with the 9-item Fear of Cancer Recurrence Inventory Short Form (FCRI-SF). Secondary outcomes include a) anxiety and depression assessed with the The Hospital Anxiety and Depression Scale (HADS), b) patient reported intervention usefulness assessed with the Patient Centered Communication Scale (PCC), c) metacognition assessed with the metacognitions questionnaire (MCQ-30), d) unmet needs assessed with Subscale of the Survivors Unmet Need Survey (SUNS-8), e) rumination assessed with the Penn State Worry Questionnaire (PSWQ), and f) General Quality of Life (QoL) assessed with the EQ-5D for later use in cost-effectiveness analysis. All measures will be completed at all three time-points (T1-T3).

At six months, the investigators will ask a subset of 15-20 patients to participate in a semi-structured phone interview about their experience with the intervention.

Oncologists:

Oncologists complete a general item on self-efficacy in managing patient FCR together with the 27-item Self-efficacy in Patient-Centeredness Questionnaire (SEPCQ-27) at baseline, post-training (only oncologists in the intervention group), and after completed inclusion. Based on a suggested framework for implementation outcomes, the investigators will assess with 11-point scales: 1) acceptability, 2) appropriateness, 3) feasibility, together with 4) fidelity, measured as the average number of components oncologists report having delivered to patients, and 5) sustainability measured as the proportion of oncologists in the intervention group who report having used CIFeR at least once within the last three months, measured six months after completed inclusion. Six months after the inclusion of their last patient, all oncologists will be asked to participate in a semi-structured interview and provide feedback on the CIFeR-training and their experiences with the intervention, including perceived utility and the perceived barriers and facilitators to implementing CIFeR in routine care. The investigators will also examine CIFeR e-training analytics regarding access and time spent on the various parts.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 18 years old
* Have completed their primary treatment, i.e., surgery, adjuvant chemotherapy, and/or radiotherapy, for breast, ovarian, prostate, or lung cancer at the participating departments between three weeks and three months previously.
* Score >= 13 on the FCRI-SF

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Fear of cancer recurrence | T1 (2 weeks prior to intervention), T2 (one week post intervention), T3 (three months post intervention)
  Assessed with the 9-item Fear of Cancer Recurrence Inventory Short Form (FCRI-SF), range 0-36. Higher scores indicate worse outcome

SECONDARY OUTCOMES:
Anxiety and depression | T1 (2 weeks prior to intervention), T2 (one week post intervention), T3 (three months post intervention)
  Assessed with the The Hospital Anxiety and Depression Scale (HADS), range 0-21. Higher scores indicate worse outcome
Patient reported intervention usefulness | T1 (2 weeks prior to intervention), T2 (one week post intervention), T3 (three months post intervention)
  Assessed with the Patient Centered Communication Scale (PCC), range 7-28. Lower scores indicate worse outcome.
Metacognition | T1 (2 weeks prior to intervention), T2 (one week post intervention), T3 (three months post intervention)
  Assessed with the metacognitions questionnaire (MCQ-30). The MCQ-30 assesses various aspects of metacognition, including subscales: cognitive confidence, positive beliefs, cognitive self-consciousness, uncontrollability and danger, and the need to control thoughts. Subscale scores range from 6 to 24. Higher scores indicate greater conviction in metacognitive beliefs.
Unmet needs | T1 (2 weeks prior to intervention), T2 (one week post intervention), T3 (three months post intervention)
  Assessed with Subscale of the Survivors Unmet Need Survey (SUNS-8), range 0-32. Higher scores indicate worse outcome.
Rumination | T1 (2 weeks prior to intervention), T2 (one week post intervention), T3 (three months post intervention)
  Assessed with the Penn State Worry Questionnaire (PSWQ), range 5-25. Higher scores indicate worse outcome.
General Quality of Life (QoL) | T1 (2 weeks prior to intervention), T2 (one week post intervention), T3 (three months post intervention)
  Assessed with the EuroQol Group Association EQ-5D-L5, representing five domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with each five severity levels. Higher levels indicate worse outcome.

OTHER OUTCOMES:
Self-efficacy (Oncologists) | At Baseline, post-training (1-3 weeks post inclusion)(only oncologists in the intervention group), and after completed inclusion of patients (time frame depends on inclusion rate).
  27-item Self-efficacy in Patient-Centeredness Questionnaire (SEPCQ-27), range 0-108. Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, Professsor, Principal Investigator — Aarhus University and Aarhus University Hospital, Denmark
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request an in accordance with the GDPR regulations
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available upon request from time of publication and 5 year post publication
Access Criteria: Written request to the primary investigator